CLINICAL TRIAL: NCT04417634
Title: Pullback wIth Resting Full-Cycle Flow ratIO or Fractional Flow Reserve for the Prediction of Post-PCI Hemodynamic Outcomes. A Study in Patients With Diffuse Coronary Artery Disease
Brief Title: RFR and FFR for the the Prediction of Post-PCI Results
Acronym: PICIO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Tommaso Gori, Clinical Professor, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-1
Record Dates: First submitted 2020-06-01; First posted 2020-06-05 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease
Keywords: stent; coronary stenosis; Angina
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Angina Pectoris

STUDY DESIGN:
Intervention Model Description: The study is a single-center, randomized superiority trial to compare two strategies for the assessment of the hemodynamic relevance of coronary lesions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RFR: resting full-cycle ratio (Experimental): RFR will be used to drive PCI
  Interventions: Diagnostic Test: RFR
- FFR: fractional flow reserve (Active Comparator): FFR will be used to drive PCI
  Interventions: Diagnostic Test: FFR

INTERVENTIONS:
Diagnostic Test: RFR — Measurement of resting flow ratio
  Arms: RFR: resting full-cycle ratio
Diagnostic Test: FFR — Measurement of fractional flow reserve
  Arms: FFR: fractional flow reserve

SUMMARY:
The aim of this study is to record hemodynamic pullback information using continuous resting full-cycle flow ratio (RFR) and fractional flow reserve (FFR) in patients with diffuse coronary artery disease. The capacity of the two indexes to predict the hemodynamic outcome after stenting will be compared.

Goals of the study are:

* To study the accuracy of RFR/FFR gradients in predicting the change in whole-vessel RFR/FFR after PCI.
* To identify a threshold in the RFR/FFR gradient that is predictive of pathological RFR/FFR also after the PCI of the first lesion.

DETAILED DESCRIPTION:
The study of the hemodynamic relevance of coronary stenoses is a well-validated method to identify coronary lesions to be treated. A number of studies show that FFR-guided PCI is superior to angiography guided PCI2-4. The achievement of maximal hyperemia is a prerequisite for FFR measurements. Hyperemia is usually achieved with the intravenous or intracoronary infusion of adenosine, which requires time and is potentially associated with discomfort for the patient. To avoid this, resting indexes have been developed. The instantaneous flow reserve (iFr) was the first of these indexes, and two large studies have shown that this parameter is non-inferior to FFR in terms of patient prognosis5. More recently, a number of other parameters have been developed, among which the RFR (resting flow ratio), which can be measured with the same intracoronary wire as the FFR and therefore requires no additional procedures. Studies show that these methods are equivalent6. The advantage of these resting indexes (which are all included in the most recent AHA/ACC guidelines7, 8), is that they do not require hyperemia. This might represent a particular advantage in the setting of tandem stenoses or diffuse disease. Since hyperemic flow in a vessel is limited by each one of the stenoses present in that vessel, each individual stenosis limits the capacity of FFR to assess the hemodynamic relevance of the other ones. In other words, invasive measurements of coronary hemodynamics using FFR in the setting of diffuse or tandem lesions are complicated by the fact that maximal hyperemia cannot be achieved, which limits the capacity of FFR to assess the hemodynamic relevance of individual focal stenoses. In this setting, the usual binary system (FFR < or > 0.80) cannot be easily applied.

This limitation is independent of the sequence of the stenoses: proximal lesions limit the reliability of FFR measurements in distal stenoses and vice versa (as long as no significant side branches are present between the two lesions). Since hyperemic flow declines significantly as soon as a 50% reduction in lumen diameter is present, even apparently non-relevant lesions may compromise any assessment based on hyperemia. This phenomenon, called hemodynamic interdependence of stenoses under conditions of hyperemia represents a significant limitation that applies to FFR but not to hyperemia-free indexes.

In order to address this issue in routine practice, FFR is measured first, then a pullback is performed and the lesion/segment where the pullback identifies the highest gradient is treated first. The removal of this stenosis increases maximal achievable hyperemic flow, thus increasing the significance of the remaining lesions. FFR is then measured again to test the hemodynamic significance of the other stenoses at a higher level of hyperemia. The capacity of FFR to predict whether removal of the first stenosis will be associated with the normalization of FFR is very limited, which requires that FFR be measured multiple times, prolonging the procedure and increasing the discomfort for the patient.

When studying coronary stenoses, the advantage of resting hemodynamic indexes is that non-critical stenoses (ie below 90%) do not modify resting blood flow. Because resting flow is more constant, and the effect of PCI is minimal, resting pressure changes measured across sequential lesions are likely to be more predictable.The hypothesis of the study is that, as compared to FFR, RFR will provide a better estimate of post-PCI hemodynamic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet ALL of the inclusion criteria:

  * Clinical indication for elective percutaneous coronary intervention of a stenosis >40% and <90% with clinical indication to percutaneous intervention (PCI) requiring functional assessment. Note: the decision to perform functional assessment will have to be taken before, and independently of, the inclusion and randomization in the study.
  * Documented heart team (when applicable, as per guidelines) decision for revascularization via PCI
  * Patient ≥18 years old

Exclusion Criteria:

* Patients will be excluded if ANY of the exclusion criteria is met:

  * Cardiogenic shock
  * Any contraindication to PCI according to guidelines
  * Presence of a coronary artery bypass grafting (CABG) in the territory under study
  * Culprit vessels in patients with ST-segment elevation myocardial infarction (STEMI)
  * TIMI (Thrombolysis in Myocardial Infarction) flow grade < 3
  * Lesion severity > 90% by visual assessment
  * Presence of thrombus
  * Participation in another randomized interventional study
  * Patient unable to give informed consent
  * Women of child-bearing potential or lactating

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-10 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Absolute difference between RFR observed and expected as compared to FFR observed versus expected. | 1 day
  Comparison of |RFRexp-RFRobs| vs. |FFRexp-FFRobs| (i.e., absolute differences between expected and observed final hemodynamic result) RFRexp and FFRexp are defined as (RFRbas plus RFRGrad) and (FFRbas plus FFRGrad)

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Cardiology, Cardiology I, university hospital Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No